CLINICAL TRIAL: NCT06182137
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation (rTMS) in The Treatment of Gambling Disorder in Indonesia: A Randomized Controlled Trial
Brief Title: Repetitive Transcranial Magnetic Stimulation (rTMS) in The Treatment of Gambling Disorder in Indonesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Kristiana Siste, Dr. dr. Kristiana Siste, SpKJ(K) - Head of Department of Psychiatry, Faculty of Medicine, Indonesia University, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KET-1499-2023
Record Dates: First submitted 2023-12-06; First posted 2023-12-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Gambling Disorder
MeSH Terms: conditions — Gambling | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- rTMS and CBT (Experimental): During 5 weeks of therapy, the subjects will undergo 12 CBT sessions combined with 15 rTMS procedures lasting about 30-60 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)
- Sham and CBT (Sham Comparator): During 5 weeks of therapy, the subjects will undergo 12 CBT sessions combined with 15 rTMS procedures (coil replaced with sham) lasting about 30-60 minutes.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — A randomised controlled trial (RCT) of 60 subjects will be conducted to evaluate the effectiveness of transmodalistic therapy with a combination of rTMS and Cognitive Behavioral Therapy (CBT) for online gambling disorder.

SUMMARY:
Research has shown that cognitive-behavioral therapy (CBT) is an effective treatment for gambling disorder. Several studies had also been done to evaluate the effectiveness of Repetitive Transcranial Magnetic Stimulation (rTMS) in addiction management, particularly in alleviating craving. A randomised controlled trial (RCT) of 30 subjects would be conducted to evaluate the effectiveness of transmodalistic therapy with a combination of rTMS and CBT for online gambling disorder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with pathological gambling (SOGS score ≥ 5)
* Subjects aged 18-59 years old
* Subjects who understand Bahasa Indonesia
* Subjects who agree to participate and receive treatment

Exclusion Criteria:

* Subjects with history of psychotic disorder, personality disorder, or sleep disorder according to ICD-11
* Subjects with history of neurostimulation
* Subjects with history of medical implant
* Subjects with history of severe neurological disorder, which causes seizure or loss of consciousness
* Subjects with intellectual disability
* Subjects with endocrinological disorders
* Subjects with contraindication during prior MR or other related procedures
* Subjects who are currently or expecting pregnancy
* Subjects with history of substance use in the last 6 months

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in pathological gambling score | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  South Oaks Gambling Screen (SOGS), Indonesian version, with minimum score of 0 and maximum score of 20. A score of 0-2 indicates no pathological gambling; a score of 3-4 indicates problems with gambling, and a score of 5 or more indicates that the subject is a probable pathological gambler. Lower score indicates a better outcome.
Improvement in gambling symptoms severity | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Gambling Symptoms Assessment Scale (G-SAS), Indonesian version, with minimum score of 0 and maximum score of 48. Interpretations: Mild (8-20), Moderate (21-30), Severe (31-40), and Extreme (41-48). Lower score indicates a better outcome.
Improvement in gambling urge | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Gambling Urge Scale (GUS), Indonesian version, with minimum score of 0 and maximum score of 42. Lower score indicates a better outcome.
Improvement in gambling related cognitive distortions | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Gambling Related Cognitions Scale (GRCS), Indonesian version, with 5 cognitive distortion domains. Lower score indicates a better outcome.

SECONDARY OUTCOMES:
Improvement in gambling-related cognitive functions | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Creyos (formerly Cambridge Brain Sciences, CBS), measures 12 domains of cognitive function with the subject results compared with their respective average age results in percentile. A higher percentile is a better outcome.
Improvement in depression symptoms | Baseline (week 0), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Beck Depression Inventory-II (BDI II), measures severity of depression symptoms, with minimum score of 0 and maximum score of 63. Interpretation: (1) minimal (0-13), (2) mild (14-19), (3) moderate (20-28), and (4) severe (29-63). Lower score indicates a better outcome.
Improvement in self-reported psychological distress | Baseline (week 0), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  20-item Self-Reporting Questionnaire (SRQ-20), Indonesian version, measures non-specific psychological distress. Score range 0-20, with scores >10 classified as mental distress. Lower score indicates a better outcome.
Improvement of overall severity of illness | Baseline (week 0), interim assessment (week 3), post-intervention (week 6), follow up at 3 months and 6 months after intervention
  Clinical Global Impression (CGI), measure overall severity of illness and improvement observed by the clinician. Lower score indicates a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Jakarta Pusat, Jakarta Special Capital Region, Indonesia